CLINICAL TRIAL: NCT04587726
Title: Dove Self-Esteem Project: Evaluating the Impact of Body Image Edutainment on Young People's Body Confidence and Self-esteem
Brief Title: Evaluating the Impact of Body Image Edutainment on Adolescent Girls' Body Image
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6423321
Record Dates: First submitted 2020-09-23; First posted 2020-10-14 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Body Image; Eating Disorder Symptom

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Girl's room video
- Control Group (Active Comparator)
  Interventions: Other: Control video - Chicken Girls

INTERVENTIONS:
Behavioral: Girl's room video — Girls Room, a body image mini-series, developed in collaboration with Lena Waithe, Dove and CAR.
  Video content was informed by empirical evidence related to body image prevention and intervention. The series consists of five, 3-minute videos.
  The videos follow the lives of a 5 best friends, and each video targets a key risk factor for body image:
  1. Appearance comparison
  2. Body appreciation
  3. Body talk
  4. Body functionality
  5. Appearance teasing & bullying
  6. Appearance focus
  The five videos aired on Instagram TV (IGTV) in March 2020.
  Arms: Intervention Group
Other: Control video - Chicken Girls — Chicken Girl's Episode - appearance neutral episode matched for target audience and video length
  Arms: Control Group

SUMMARY:
Body image is one of the leading concerns for young people. These concerns may can have serious consequences, including anxiety, depression, risk taking behaviours, eating disorders and suicidal ideation.

An extensive body of research highlights the negative effects associated with viewing idealistic media among adolescents. More recently, research has looked at harnessing media and technology to develop and disseminate material that counteracts these harmful effects. Using 'edutainment' (entertainment with educational content) to develop and disseminate interventions is a novel avenue of research. Micro-interventions (brief, low intensity, self-administered interventions), offer an alternative to traditional, intense interventions that may be unsuitable for milder concerns. Body image micro-interventions have proven effective at providing immediate and short-term improvements in body image among women. To date, body image micro-interventions have been focused on adult samples, with little research exploring how this intervention model may cater to adolescents.

The aim of the present study is to conduct a randomised controlled trial to evaluate the efficacy of a brief body image video micro-intervention to improve body image and acceptance of appearance diversity among girls, in addition to appearance-related internalised racism among the Black subgroup of girls.

The body image video micro-intervention is a 3-minute episode from Girls Room; a mini-series developed to address risk factors for body image. The series was developed through a collaboration between Lena Waithe, Dove (Unilever) and the Centre for Appearance.

The comparison control group will watch a 3-minute episode from an equivalent popular series which does not contain any appearance-related content.

In addition to the outcomes of interest, post-video acceptability checks will also be assessed to determine viewers' enjoyment, engagement, and identification with the video, as well as their intent to re-engage and share.

To undertake this project, 1848 adolescent girls will be recruited via an external research agency. Female-identifying North American citizens, aged 12-18 years old will be recruited, stratified to include 50% Black and 50% non-Black adolescents. The participants will be randomised to watch either the Girls Room episode, or control episode, at either 25%, 50% or 100% length of exposure. Before watching the video, they will complete baseline measures of demographics, state body satisfaction, acceptance of diversity of appearance, and appearance-related internalised racism (Black girls only). They will then be exposed to the video, before completing the measures again (post-exposure), along with acceptability checks. Participants will then be provided with a debrief of study aims and a list of support sources.

DETAILED DESCRIPTION:
Background

Body image is one of the leading concerns for young people. This is particularly concerning, given that body dissatisfaction is a key risk factor for serious mental and physical health issues, including anxiety, depression, risk taking behaviours, eating disorders and suicidal ideation.

An extensive body of research highlights the negative effects associated with viewing idealistic media among adolescents. More recently, research has looked at harnessing media and technology to develop and disseminate material that disrupts and counteracts these harmful effects. 'Edutainment', entertainment with educational content, is an effective method for delivering and modelling health promotion material in mainstream media. Further, it offers an alternative to traditional, intense interventions that are, at times, unnecessary or unsuitable for milder concerns.

Body image micro-interventions have proven effective at providing immediate and short-term improvements in body image among adult women, and research is beginning to explore their impact among young people. A recent study found that evidence-informed body image animations produced immediate and short-term improvements in children's body satisfaction, media literacy, and self-efficacy in addressing appearance teasing. However, these effects were less potent for older children (i.e., adolescents); which may be attributable to the use of cartoons, as opposed to real-life characters. The effects of viewing real-world depictions of positive body image attitudes and behaviours has yet to be evaluated.

In collaboration with Dove (Unilever) and Lena Waithe (an Emmy-Award winning American screenwriter, producer and actress), body image experts from the Centre for Appearance Research (CAR) developed a series of brief videos that depict real-life characters addressing key risk factors for body image concerns.

This study aims to evaluate the acceptability and impact of viewing one 5-minute episode of Girls Room (Episode 1: One of One') on the body image of 13-18-year-old girls from the US. The research questions are as follows:

1. Does watching Girls Room result in improved body image and acceptance of diversity of appearance among adolescent girls compared with watching an equivalent series that is popular among adolescent girls and typical of content on Instagram?

a. Are these effects moderated by the ethnicity of the viewer (Black versus all other ethnicities)?

3. Does watching Girls Room result in reduced appearance-related internalized racism among Black adolescent girls compared with watching an equivalent series that is popular and typical of content on Instagram?

Design

This study adopts an experimental pre-post 2 x 2 design, which includes following two independent variables:

1. Ethnicity of viewer (2 Levels) i. Black ii. Non-Black (this will include all other ethnicities expect Black)
2. Video condition (2 levels) i. Body image video (Girls Room) ii. Equivalent series that is popular among adolescent girls and typical of content on Instagram (Chicken Girls)

There are three outcome measures (dependent variables) of interest:

1. State Body Image (primary outcome)
2. State Acceptance of Diversity of Appearance (secondary outcome)
3. State Appearance-related Internalized Racism- to be measured among Black girls only (secondary outcome)

There is also one moderator:

1. Ethnicity of the viewer (Black vs. Non-Black)

Participants & Recruitment

The current content is aimed at improving body image risk factors and increasing knowledge and protective factors prevalent amongst adolescent girls. Therefore, the research will utilise a representative sample of North American girls aged 12-18 years old. They will be stratified to be 50% Black and 50% other ethnicities, who are current users of Instagram or YouTube.

To achieve the agreed upon research objectives and in alignment with project timelines, the recruitment process will be out-sourced to an external professional recruitment agency. The agency's brief will outline the following inclusion criteria; female North American citizens, aged 12-18 years old; English speaking, not participated in academic or market research elated to mental health or social media in the preceding 6 months. Participants will be offered agency credit for their participation.

A sample size of 640 (160 girls per cell) is necessary for 80% power to detect a partial eta squared as low as 0.012, and based on the assumption that there will be a correlation between Time 1 (pre) and Time 2 (post) measures of 0.5.

Intervention

Girls Room, a body image mini-series, was developed in collaboration with Lena Waithe, Dove and CAR. Video content was informed by empirical evidence related to body image prevention and intervention. The series consists of five, 3-minute videos, with each video targeting a key risk factor for body image (see below). The five videos aired on Instagram TV (IGTV) in March 2020.

Procedure

Girls will not be briefed on the purpose of the study, the research questions, or their condition prior to or during study participation. However, they will be given sufficient information to provide informed consent. They will also be advised that they may be asked the same questions twice throughout the study. After completing the study, participants should be fully debriefed and provided with sources of support.

The online study will include validated, age-appropriate, self-report measures that assess demographics and the immediate impact of video exposure on adolescents' body image and associated risk and protective factors. Outcome assessments will be conducted at two time points, including immediately before (time one) and after video exposure (time two). Assessments and video exposure will occur within one session. The survey will be conducted online, at home, and should take no longer than 25 minutes for participants to complete.

Recruitment and survey dissemination will be conducted by a third-party research agency. The agency will contact eligible participants via their parents, with consent required by both parent and child. Following consent, the child will participate in a once-off survey that consists of four phases:

1. Baseline assessments of demographics, body image, acceptance of appearance diversity, internalised racism (Black participants only)
2. Randomisation into exposure condition
3. Video exposure
4. Post-exposure assessments of body image, acceptance of appearance diversity, internalised racism (Black participants only), acceptability checks (Enjoyment, Engagement, and Identification, Re-engagement, and Sharing)

Participants will then be provided with a debrief of study aims and a list of support sources.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and literate
* Instagram/You Tube users
* 12-18 years
* Female north American citizens
* Not participated in academic or market research related to mental health or social media in the preceding 6 months

Exclusion Criteria:

* Not Instagram/YouTube users
* Identify as male
* Outside US
* No access to internet/online
* Participated in academic or market research related to mental health or social media in the past 6 months

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Identify as female
Enrollment: 686 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Change in State body satisfaction | Immediately pre-intervention and immediately post-intervention (change)
  Measured via Visual Analogue Scales (Richardson & Paxton, 2010; McLean, Paxton & Wetherheim, 2016). 6-items for the measure, VAS scales (min 0 max 100), along with 12 filler items and 4 attention checks.

SECONDARY OUTCOMES:
Change in Acceptance of appearance diversity | Immediately pre-intervention and immediately post-intervention (change)
  Adapted measure (based on Masnari et al., 2013; Parnell et al., under review; Matheson et al., in press). 4 different characters are shown, with 9-items for each presented on a VAS scale (opposite anchors e.g. mean-nice, sad-happy, unpopular-popular) , as well as attention checks throughout (every 3 items).
Change in Internalised Racism (Black sample only) | Immediately pre-intervention and immediately post-intervention (change)
  Measured via VAS scales adapted from the Alteration of Physical Appearance (APA) and Hair Change (HC) subscales of the Internalized Racial Oppression Scale for Black Individuals (Bailey et al., 2011). 3 of the 8 items are removed as they refer to behaviours/perceptions of others, rather than attitudes about their own appearance. Attention checks are included every 4th item
Intervention acceptability | Immediately post-intervention
  Measured on 12 VAS scales (min 0, max 100), assessing enjoyment, engagement, identification, and intent to re-engage and share. 2 attention checks are included.

CONTACTS AND LOCATIONS:
Locations (1):
- MetrixLab, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No